CLINICAL TRIAL: NCT03445026
Title: Frequency of Hypodontia After Chemotherapy in Childhood Cancer Survivors: A Cross Sectional Study
Brief Title: Frequency of Hypodontia After Chemotherapy in Childhood Cancer Survivors Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Adel Mahmoud, B.D.Sc,MFDS RCSEd,Dentist at 57357 Children Cancer Hospital, Cairo University
Other Study IDs: CEBD-CU-2018-02-20
Record Dates: First submitted 2018-02-20; First posted 2018-02-26 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Hypodontia
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: dental panorama — radiographic examination

SUMMARY:
This study aims to provide information on the frequency of hypodontia in children cancer survivors receiving chemotherapy before 4 years of age.Patients who met the eligibility criteria will be given a structured questionnaire to fill followed by a radiographic examination (dental panorama) for confirmation and standardization of the results.

ELIGIBILITY:
Inclusion Criteria:

* Aged 4 years or less when they first started their antineoplastic chemotherapy
* Both genders
* Able to cooperate

Exclusion Criteria:

* Children with known family history of hypodontia
* Children with any associated developmental anomalies (eg, ectodermal dysplasia, cleft lip or palate and Down syndrome)
* Children who received radiotherapy
* Children with previous loss of teeth due to trauma, caries, periodontal disease or extraction 5- Children who received bone marrow transplantation 6-Parents/patients unwilling to give informed consent

Min Age: 6 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be selected from 57357 Children Cancer Hospital records according to inclusion and exclusion criteria and contacted to attend.
Sampling Method: Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Hypodontia | 1 year
  missing not formed teeth

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
BDS,MFDS RCSEd Dentist at 57357 Children Cancer Hospital Egypt